CLINICAL TRIAL: NCT03083847
Title: Sanaria PfSPZ Challenge With Pyrimethamine Chemoprophylaxis (PfSPZ-CVac Approach): Phase 1 Dose Escalation Trial to Determine Safety and Development of Protective Efficacy After Exposure to Only Pre-erythrocytic Stages of Plasmodium Falciparum
Brief Title: Dose Escalation PfSPZ-CVac
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Sanaria Inc. (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 170067; 17-I-0067
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Results first posted 2020-07-24 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2019-12-09

CONDITIONS: Malaria
Keywords: Malaria; Parasitemia; Immune; Responses; Sporozoites
MeSH Terms: conditions — Malaria; Parasitemia | interventions — chloroquine diphosphate; Pyrimethamine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Pilot (1a): 1 injection of 5x10^4 PfSPZ Challenge+pyrimethamine (Experimental): Pilot Phase - 1 injection of 5x10^4 sporozoites of PfSPZ Challenge (NF54) with 50mg of pyrimethamine dosed on days 2 and 3 after injection
  Interventions: Drug: Pyrimethamine; Biological: Sanaria PfSPZ Challenge
- Pilot (1b):1 injection of 1x10^5 PfSPZ Challenge+pyrimethamine (Experimental): Pilot Phase - 1 injection of 1x10^5 sporozoites of PfSPZ Challenge (NF54) with 50mg of pyrimethamine dosed on days 2 and 3 after injection
  Interventions: Drug: Pyrimethamine; Biological: Sanaria PfSPZ Challenge
- Pilot (1d):1 injection of 2x10^5 PfSPZ Challenge+pyrimethamine (Experimental): Pilot Phase - 1 injection of 2x10^5 sporozoites of PfSPZ Challenge (NF54) with 50mg of pyrimethamine dosed on days 2 and 3 after injection
  Interventions: Drug: Pyrimethamine; Biological: Sanaria PfSPZ Challenge
- Pilot (5a): 1 injection of 1x10^5 PfSPZ Challenge+chloroquine (Experimental): Pilot Phase - 1 injection of 1x10^5 sporozoites of PfSPZ Challenge (NF54) with 1000mg of chloroquine (loading dose) 2 days prior to injections and 500mg (maintenance dose) 5 days post injection
  Interventions: Drug: Chloroquine Phosphate; Biological: Sanaria PfSPZ Challenge
- Pilot (5b): 1 injection of 2x10^5 PfSPZ Challenge+chloroquine (Experimental): Pilot Phase - 1 injection of 2x10^5 sporozoites of PfSPZ Challenge (NF54) with 1000mg of chloroquine (loading dose) 2 days prior to injections and 500mg (maintenance dose) 5 days post injection
  Interventions: Drug: Chloroquine Phosphate; Biological: Sanaria PfSPZ Challenge
- Main (2a):3 doses of 2x10^5 PfSPZ Challenge+pyrimethamine+NF54 (Experimental): Main Phase - 3 monthly doses of 2x10^5 sporozoites of PfSPZ Challenge + pyrimethamine on days 2 and 3 post injection + homologous controlled human malaria infection (CHMI) with 3.2x10^3 PfSPZ Challenge (NF54) at 12 weeks after third injection
  Interventions: Drug: Pyrimethamine; Biological: Sanaria PfSPZ Challenge
- Main (2b):3 doses of 2x10^5 PfSPZ Challenge+pyrimethamine+7G8 (Experimental): Main Phase - 3 monthly doses of 2x10^5 sporozoites of PfSPZ Challenge + pyrimethamine on days 2 and 3 post injection + heterologous CHMI with 3.2x10^3 PfSPZ Challenge (7G8) at 12 weeks after third injection
  Interventions: Drug: Pyrimethamine; Biological: Sanaria PfSPZ Challenge
- Main (3):3 doses of 2x10^5 PfSPZ Challenge+chloroquine+7G8 (Experimental): Main Phase - 3 monthly doses of 2x10^5 sporozoites of PfSPZ Challenge + weekly chloroquine (1000mg given 2 days prior to injections and 500mg given 5 days post injection and weekly thereafter until 5 days post third injection) + heterologous controlled human malaria infection (CHMI) with 3.2x10^3 PfSPZ Challenge (7G8) at 12 weeks after third injection
  Interventions: Drug: Chloroquine Phosphate; Biological: Sanaria PfSPZ Challenge
- Main Phase (4a) - Infectivity Control: NF54 (homologous) CHMI (Experimental): Main Phase - Infectivity Control with one dose of 3.2x10^3 sporozoites of PfSPZ Challenge (NF54) (homologous) controlled human malaria infection (CHMI)
  Interventions: Biological: Sanaria PfSPZ Challenge
- Main Phase (4b) - Infectivity Control: 7G8 (heterologous) CHMI (Experimental): Main Phase - Infectivity Control with 3.2x10^3 sporozoites of PfSPZ Challenge 7G8 (heterologous) controlled human malaria infection (CHMI)
  Interventions: Biological: Sanaria PfSPZ Challenge

INTERVENTIONS:
Drug: Chloroquine Phosphate — Chloroquine has been widely used for treatment and prophylaxis of malaria since 1946 (Most, London et al. 1984). It was the treatment of choice for uncomplicated malaria for decades because it was safe, well tolerated, affordable and highly effective for the treatment of malaria. However, increasing spread of chloroquine- resistant Pf over the last two decades has severely limited its use (Wellems 2002). Chloroquine phosphate is U.S Food and Drug Administration (FDA) approved for suppressive treatment (prophylaxis) and for acute attacks of malaria due to P. vivax, P. malariae, P. ovale, and susceptible strains of Pf.
  Arms: Main (3):3 doses of 2x10^5 PfSPZ Challenge+chloroquine+7G8; Pilot (5a): 1 injection of 1x10^5 PfSPZ Challenge+chloroquine; Pilot (5b): 1 injection of 2x10^5 PfSPZ Challenge+chloroquine
Drug: Pyrimethamine — Pyrimethamine is a folic acid antagonist that has been commonly used as antimalarial drug for both treatment and prevention of malaria, usually in combination with sulfadoxine in adults, pregnant women, and children worldwide (Organization April 2013 (rev. January2014)
  Arms: Main (2a):3 doses of 2x10^5 PfSPZ Challenge+pyrimethamine+NF54; Main (2b):3 doses of 2x10^5 PfSPZ Challenge+pyrimethamine+7G8; Pilot (1a): 1 injection of 5x10^4 PfSPZ Challenge+pyrimethamine; Pilot (1b):1 injection of 1x10^5 PfSPZ Challenge+pyrimethamine; Pilot (1d):1 injection of 2x10^5 PfSPZ Challenge+pyrimethamine
Biological: Sanaria PfSPZ Challenge — Sanaria Inc has manufactured two strains of Sanaria PfSPZ Challenge: NF54 and 7G8. The Sanaria PfSPZ Challenge contains fully infectious PfSPZ purified from the salivary glands of Anopheles stephensi mosquitoes raised under aseptic conditions. The infectious PfSPZ are formulated in cryoprotectant to maintain potency for an extended period. Sanaria PfSPZ Challenge (NF54) is known to be susceptible to chloroquine, pyrimethamine, atovaquone, artesunate, but not mefloquine. Sanaria PfSPZ Challenge (7G8) is known to be susceptible to mefloquine, atovaquone, artemether and artesunate but not to chloroquine or pyrimethamine.

SUMMARY:
Background:

People get malaria from bites from infected mosquitos. Researchers are studying a vaccine strategy. They will give people malaria parasites by injecting them with live infectious malaria parasites with antimalarial medications and then see if this strategy prevents malaria infection while off antimalarial medications.

Objective:

To see if combining a high dose of live, infectious malaria parasites (known as Sanaria PfSPZ Challenge) and two FDA approved drugs that kill malaria parasites (pyrimethamine [PYR] OR chloroquine [CQ]) is safe and can provide people protection against malaria.

Eligibility:

Healthy adults ages 18-50 who:

* are not pregnant or breastfeeding or planning on becoming pregnant while in the study
* are not infected with HIV, Hepatitis B or Hepatitis C
* have reliable early morning access to the NIH Clinical Center
* are able to come to the outpatient clinic frequently, sometimes daily
* have not been diagnosed with malaria within the past 10 years

Design:

* Participants will be screened with medical history and physical exam. They will have heart, blood, and urine tests.
* Participants will have blood drawn for tests at most visits.
* Participants will keep track of their temperature and symptoms during some sections of the study.
* Participants will join one part of the study.

Part 1 is one month:

* Participants will get the parasites by an injection into a vein on day 1 and receive antimalarial medications.
* They will have daily visits on days 7-14
* They will take another antimalarial at visits on days 15-17.
* The final visit will be on day 29.

Part 2 is seven months:

* For the first 3 months, participants will get the parasite injection into a vein for 3 injections in total. Each injection will occur once per month while taking an antimalarial drug.
* They will have daily visits on days 7-14 after the first injection, and on days 7-11 after the second and third injection.
* They will have a final (fourth) injection around month 6 without any antimalarial medication.
* After this fourth injection, participants may have up to 21 daily visits from day 7 after injection until end of study.

Part 3 is one month:

* Participants will get the parasites by injection into a vein on day 1 without antimalarial medications.
* They will have visits almost every day starting day 7 from injection.
* They will take an antimalarial medication when they are diagnosed with malaria
* They will return for final end of study visit on days 27-29.

DETAILED DESCRIPTION:
Human studies have shown that immunization by the bite Plasmodium falciparum (Pf) sporozoite(SPZ)-infected mosquitoes under drug coverage with chloroquine, an approach called chemoprophylaxis with sporozoites (CPS) or infection treatment vaccination (ITV), can provide high level, long term protection against homologous controlled human malaria infection (CHMI). The Sanaria PfSPZ chemoprophylaxis vaccination (PfSPZ CVac) approach duplicates this with an injectable SPZ regimen. In both approaches, whether mosquitoes or syringes are used for SPZ administration, when chloroquine is used as the chemoprophylactic agent, transient, limited, asexual erythrocytic stage is seen in the majority of participants. Thus the question remains whether the significant protective efficacy seen can be achieved with pre-erythrocytic (sporozoite/liver stage) exposure only.

Previously, we performed a phase 1 study to investigate the safety, tolerability, immunogenicity, and protective efficacy of Sanaria PfSPZ CVac with chloroquine (sporozoites, liver, and blood stage) or pyrimethamine with chloroquine (sporozoites and liver stage only) to further describe stage specific sterile protection (NIAID protocol #15-I-0169). In this study, we demonstrated that pyrimethamine is safe to administer, well tolerated, and can prevent subpatent and patent parasitemia (qPCR and blood smear negative) 100% of the time during Sanaria PfSPZ CVac. The study also duplicated the results previously reported with Sanaria PfSPZ CVac with chloroquine in terms of safety profile and protective efficacy against homologous CHMI. Although a combination of Sanaria PfSPZ- CVac with pyrimethamine and PfSPZ Challenge at 51,200 PfSPZ did not provide a significant protection level against homologous CHMI, we demonstrated that some subjects did develop protective immunity without any evidence of blood stage exposure during PfSPZ-CVac.

Building on these results and taking the lessons learned from other pre-erythrocytic vaccine studies and models that have shown the importance of reaching a minimal antigen threshold required for the development of sterile immunity, this proposed study will assess the safety, tolerability, immunogenicity, and protective efficacy of increasing the dose of Sanaria PfSPZ Challenge sporozoites while receiving the same, or, if needed to successfully prevent parasitemia, a higher dose of pyrimethamine. Unlike the first study, however, pyrimethamine will be administered by itself as the partner drug, and will not be co-administered with chloroquine. The efficacy of PfSPZ-CVac with pyrimethamine will be assessed against CHMI with homologous parasites (Arm 2a) and CHMI with heterologous parasites (Arm 2b). Additionally, we will explore the impact of increasing the dose of Sanaria PfSPZ Challenge sporozoites while receiving chloroquine alone prophylaxis. The efficacy of PfSPZ-CVac with chloroquine will be assessed only against CHMI with heterologous parasites (Arm 3), as protection against homologous parasites has now been shown in two separate trials. It will thus be possible to compare the efficacy of the two partner drugs against heterologous CHMI. The results of this study will contribute to understanding the targets and mechanisms of immunity against Pf malaria infection and how the degree of exposure to the parasite (pre-erythrocytic or erythrocytic stage only or both) impacts these responses and subsequent protective efficacy.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal to 18 and less than or equal to 50 years.
* In good general health and without clinically significant medical history
* Malaria comprehension exam completed, passed (a score of greater than or equal to 80% or per investigator s discretion) and reviewed prior to enrollment
* Reliable access to the clinical trial center and availability to participate for duration of study
* Females of childbearing potential must be willing to use reliable contraception (as defined below) from 21 days prior to study day -2 to 28 days following last Sanaria PfSPZ Challenge exposure
* Subject to the judgment and discretion of the PI, female participants who meet ANY ONE of the criteria listed immediately below, may not be required to take any additional measures to avoid pregnancy. Such participants will be counseled on risks at the time of consent and at appropriate points (e.g. when pregnancy testing occurs) during the study:

  * Females who have had their uterus, and/or BOTH ovaries removed
  * Females who have had BOTH fallopian tubes surgically 'tied' or removed
  * Females who are above the age of 45 and have spontaneously had no menses at any point during the past 12 or more consecutive months (i.e. have reached menopause)
  * Females who, in the conservative and reasonable judgment of the PI (e.g. due to sexual orientation or serious life choice (such as being celibate clergy or transgender), during the entire trial will NOT participate in any potentially reproductive sexual contact
  * Females who, in the conservative and reasonable judgment of the PI, are in a monogamous stable relationship with a male who has undergone vasectomy at least 4 months prior or another procedure/medical condition that deems the male sterile
* Subject to the judgment and discretion of the PI, female participants who DO NOT meet ANY of the criteria listed above, will be appropriately counseled on reproductive risks and pregnancy avoidance, and will be required to adhere to the following measures and agree to 2 methods of pregnancy prevention as noted below:

  * CATEGORY 1: a highly effective hormonal method to prevent pregnancy [e.g. CONSISTENT, CONTINUOUS use of contraceptive pill, patch, ring, implant or injection], and/or IUD or equivalent
  * IN ADDITION TO CATEGORY 2: a barrier method to be used at the time of potentially reproductive sexual activity (e.g. [male/female condom, 'cap,' or diaphragm] + spermicide).

EXCLUSION CRITERIA:

* Currently is breast-feeding (if female).
* Pregnancy as determined by a positive urine or serum human choriogonadotropin (beta- hCG) test at any point during the study (if female).
* Recent travel to a malaria endemic area within 5 years of enrollment (Endemic areas are defined per the CDC website. Factors such as but not limited to use of antimalaria prophylaxis during travel, length of stay, activities during the travel, history of illnesses within 30 days of travel will be considered to determine the likelihood that the subject was exposed to malaria)
* Planned travel to a malaria endemic area (as defined by the Center for Disease Control) during the study period
* Reported history of confirmed malaria diagnosis on peripheral blood smear or by clinical history in the past 10 years.
* Hemoglobin, WBC, platelets, ALT, and creatinine outside of local lab normal range (subjects may be included at the investigator s discretion for not clinically significant values outside of normal range)
* Abnormal urinalysis as defined by positive urine glucose, protein, and red blood cells. Subject can be included if investigator determine the abnormality is not clinically significant .
* BMI < 17 or BMI > 35
* Anticipated use during the study period, or use within the following periods prior to enrollment:

  * Investigational malaria vaccine within the last five years
  * Malaria chemoprophylaxis within 6 months
  * Chronic systemic immunosuppressive medications (>14 days) within 6 months (e.g.cytotoxic medications, oral/parental corticosteroids >0.5 mg/kg/day prednisone or equivalent). Corticosteroid nasal spray for allergic rhinitis and topical corticosteroids for mild, uncomplicated dermatitis are allowed.
  * Blood products or immunoglobulins within 6 months
  * Systemic antibiotics with antimalarial effects within 30 days (such as clindamycin, doxycycline)
  * Investigational or non-registered product or vaccine within 30 days
  * Receipt of a live vaccine within 28 days or a killed vaccine within the 14 days prior to Sanaria PfSPZ Challenge
  * Medications known to interact with pyrimethamine and/or chloroquine (for the main and pilot study participants ONLY), atovaquone, proguanil (ALL participants)
* Reported history of:

  * Sickle cell disease, sickle cell trait, or other hemoglobinopathies
  * Splenectomy or functional asplenia
  * Systemic anaphylaxis
  * Any allergic reactions to study drugs (pyrimethamine, chloroquine) or NSAIDs, atovaquone, proguanil
  * Documented history of chronic or active neurologic disease (including seizures, uncontrolled migraine headaches)
  * Psoriasis or porphyria
  * Ocular diseases including retinopathy or visual field defects
* Clinically significant medical condition, physical examination findings, other clinically significant abnormal laboratory results, or past medical history that may have clinically significant implications for current health status and participation in the study in the opinion of the Investigator. A clinically significant condition or process includes but is not limited to:

  * A process that would affect the immune response, or requires medication that affects the immune response
  * Any contraindication to repeated phlebotomy
  * A condition or process in which signs or symptoms could be confused with reactions to malaria challenge and/or infection, including dermatologic abnormalities at the site of sporozoite inoculation
  * A chronic or subclinical condition which could be exacerbated by administration of any of the PfSPZ-CVac components or malaria infection
* History of, or known active cardiac disease including: (1) prior myocardial infarction (heart attack); (2) angina pectoris; (3) congestive heart failure; (4) valvular heart disease; (5) cardiomyopathy; (6) pericarditis; (7) stroke or transient ischemic attack; (8) exertional chest pain or shortness of breath; or ( 9) other heart conditions under the care of a doctor
* Clinically significant ECG findings, as determined by the expert study cardiologist
* Moderate or high risk for coronary heart disease (CHD) based on NHANES I cardiovascular risk assessment
* Acute illness at the time of enrollment
* Infection with HIV, Hepatitis B, Hepatitis C
* Psychiatric condition that precludes compliance with the protocol including but not limited to:

  * Psychosis within the past 3 years
  * Ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years
* Suspected or known current alcohol or drug abuse as defined by the American Psychiatric Association in the DSM V at the discretion of the PI
* Clinical trial staff and/or Sanaria Inc. employees with direct involvement in the conduct of the trial are excluded from participation.
* Participating in other clinical trials involving investigational interventions or off label medication use during the study period (excluding participation in the optional long term follow up visits). Participation in other trials such as observational or imaging studies will be discussed with the investigators.
* Any other finding that, in the judgment of the Investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a subject s ability to give informed consent, or increase the risk of having an adverse outcome from participating in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick E Duffy, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bijker EM, Borrmann S, Kappe SH, Mordmuller B, Sack BK, Khan SM. Novel approaches to whole sporozoite vaccination against malaria. Vaccine. 2015 Dec 22;33(52):7462-8. doi: 10.1016/j.vaccine.2015.09.095. Epub 2015 Oct 23. PMID 26469716
- [Background] Mordmuller B, Supan C, Sim KL, Gomez-Perez GP, Ospina Salazar CL, Held J, Bolte S, Esen M, Tschan S, Joanny F, Lamsfus Calle C, Lohr SJ, Lalremruata A, Gunasekera A, James ER, Billingsley PF, Richman A, Chakravarty S, Legarda A, Munoz J, Antonijoan RM, Ballester MR, Hoffman SL, Alonso PL, Kremsner PG. Direct venous inoculation of Plasmodium falciparum sporozoites for controlled human malaria infection: a dose-finding trial in two centres. Malar J. 2015 Mar 18;14:117. doi: 10.1186/s12936-015-0628-0. PMID 25889522
- [Background] Roestenberg M, McCall M, Hopman J, Wiersma J, Luty AJ, van Gemert GJ, van de Vegte-Bolmer M, van Schaijk B, Teelen K, Arens T, Spaarman L, de Mast Q, Roeffen W, Snounou G, Renia L, van der Ven A, Hermsen CC, Sauerwein R. Protection against a malaria challenge by sporozoite inoculation. N Engl J Med. 2009 Jul 30;361(5):468-77. doi: 10.1056/NEJMoa0805832. PMID 19641203
- [Derived] Mwakingwe-Omari A, Healy SA, Lane J, Cook DM, Kalhori S, Wyatt C, Kolluri A, Marte-Salcedo O, Imeru A, Nason M, Ding LK, Decederfelt H, Duan J, Neal J, Raiten J, Lee G, Hume JCC, Jeon JE, Ikpeama I, Kc N, Chakravarty S, Murshedkar T, Church LWP, Manoj A, Gunasekera A, Anderson C, Murphy SC, March S, Bhatia SN, James ER, Billingsley PF, Sim BKL, Richie TL, Zaidi I, Hoffman SL, Duffy PE. Two chemoattenuated PfSPZ malaria vaccines induce sterile hepatic immunity. Nature. 2021 Jul;595(7866):289-294. doi: 10.1038/s41586-021-03684-z. Epub 2021 Jun 30. PMID 34194041
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-I-0067.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Contingency arms for a higher PYR dose (75mg instead of 50mg) were not enrolled as criteria were not met for their inclusion (50mg of PYR prevented detectable parasitemia in all enrolled arms). The PYR contingency arms that were not enrolled were labelled 1c, 1e, and 1f in the protocol.
Pre-assignment Details: 121 participants were screened; 55 participants were assigned to an arm; 66 participants did not meet screening criteria; one subject was consented to two arms, but started on only a control arm.
  Participants in each Pilot phase were independent; no participant was enrolled in more than one arm or period in either the pilot or main phases.
Groups:
- Pilot (1a):1 Injection of 5x10^4 PfSPZ Challenge+Pyrimethamine: Pilot Phase - 1 injection of 5x10^4 sporozoites of PfSPZ Challenge (NF54) with 50mg of pyrimethamine dosed on days 2 and 3 after injection
Period: Pilot 1a
Arm/Group | Pilot (1a):1 Injection of 5x10^4 PfSPZ Challenge+Pyrimethamine | Pilot (1b):1 Injection of 1x10^5 PfSPZ Challenge+Pyrimethamine | Pilot (5a): 1 Injection of 1x10^5 PfSPZ Challenge+Chloroquine | Pilot (1d):1 Injection of 2x10^5 PfSPZ Challenge+Pyrimethamine | Pilot (5b): 1 Injection of 2x10^5 PfSPZ Challenge+Chloroquine | Main (2a):3 Doses of 2x10^5 PfSPZ Challenge+Pyrimethamine+NF54 | Main (2b):3 Doses of 2x10^5 PfSPZ Challenge+Pyrimethamine+7G8 | Main (3):3 Doses of 2x10^5 PfSPZ Challenge+Chloroquine+7G8 | Main Phase (4a) - Infectivity Control: NF54 (Homologous) CHMI | Main Phase (4b) - Infectivity Control: 7G8 (Heterologous) CHMI
Started | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Pilot Ib & 5a
Arm/Group | Pilot (1a):1 Injection of 5x10^4 PfSPZ Challenge+Pyrimethamine | Pilot (1b):1 Injection of 1x10^5 PfSPZ Challenge+Pyrimethamine | Pilot (5a): 1 Injection of 1x10^5 PfSPZ Challenge+Chloroquine | Pilot (1d):1 Injection of 2x10^5 PfSPZ Challenge+Pyrimethamine | Pilot (5b): 1 Injection of 2x10^5 PfSPZ Challenge+Chloroquine | Main (2a):3 Doses of 2x10^5 PfSPZ Challenge+Pyrimethamine+NF54 | Main (2b):3 Doses of 2x10^5 PfSPZ Challenge+Pyrimethamine+7G8 | Main (3):3 Doses of 2x10^5 PfSPZ Challenge+Chloroquine+7G8 | Main Phase (4a) - Infectivity Control: NF54 (Homologous) CHMI | Main Phase (4b) - Infectivity Control: 7G8 (Heterologous) CHMI
Started | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Pilot 1d & 5b
Arm/Group | Pilot (1a):1 Injection of 5x10^4 PfSPZ Challenge+Pyrimethamine | Pilot (1b):1 Injection of 1x10^5 PfSPZ Challenge+Pyrimethamine | Pilot (5a): 1 Injection of 1x10^5 PfSPZ Challenge+Chloroquine | Pilot (1d):1 Injection of 2x10^5 PfSPZ Challenge+Pyrimethamine | Pilot (5b): 1 Injection of 2x10^5 PfSPZ Challenge+Chloroquine | Main (2a):3 Doses of 2x10^5 PfSPZ Challenge+Pyrimethamine+NF54 | Main (2b):3 Doses of 2x10^5 PfSPZ Challenge+Pyrimethamine+7G8 | Main (3):3 Doses of 2x10^5 PfSPZ Challenge+Chloroquine+7G8 | Main Phase (4a) - Infectivity Control: NF54 (Homologous) CHMI | Main Phase (4b) - Infectivity Control: 7G8 (Heterologous) CHMI
Started | 0 | 0 | 0 | 4 | 4 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 4 | 4 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Main
Arm/Group | Pilot (1a):1 Injection of 5x10^4 PfSPZ Challenge+Pyrimethamine | Pilot (1b):1 Injection of 1x10^5 PfSPZ Challenge+Pyrimethamine | Pilot (5a): 1 Injection of 1x10^5 PfSPZ Challenge+Chloroquine | Pilot (1d):1 Injection of 2x10^5 PfSPZ Challenge+Pyrimethamine | Pilot (5b): 1 Injection of 2x10^5 PfSPZ Challenge+Chloroquine | Main (2a):3 Doses of 2x10^5 PfSPZ Challenge+Pyrimethamine+NF54 | Main (2b):3 Doses of 2x10^5 PfSPZ Challenge+Pyrimethamine+7G8 | Main (3):3 Doses of 2x10^5 PfSPZ Challenge+Chloroquine+7G8 | Main Phase (4a) - Infectivity Control: NF54 (Homologous) CHMI | Main Phase (4b) - Infectivity Control: 7G8 (Heterologous) CHMI
Started | 0 | 0 | 0 | 0 | 0 | 9 | 10 | 10 | 4 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 8 | 9 | 6 | 4 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Main (2a):3 Doses of 2x10^5 PfSPZ Challenge+Pyrimethamine+NF54 | Main (2b):3 Doses of 2x10^5 PfSPZ Challenge+Pyrimethamine+7G8 | Main (3):3 Doses of 2x10^5 PfSPZ Challenge+Chloroquine+7G8 | Main Phase (4a) - Infectivity Control: NF54 (Homologous) CHMI | Main Phase (4b) - Infectivity Control: 7G8 (Heterologous) CHMI | Pilot (1a):1 Injection of 5x10^4 PfSPZ Challenge+Pyrimethamine | Pilot (1b):1 Injection of 1x10^5 PfSPZ Challenge+Pyrimethamine | Pilot (1d):1 Injection of 2x10^5 PfSPZ Challenge+Pyrimethamine | Pilot (5a): 1 Injection of 1x10^5 PfSPZ Challenge+Chloroquine | Pilot (5b): 1 Injection of 2x10^5 PfSPZ Challenge+Chloroquine | Total
Number analyzed (Participants) | 9 | 10 | 10 | 4 | 8 | 2 | 2 | 4 | 2 | 4 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 10 | 4 | 8 | 2 | 2 | 4 | 2 | 4 | 55
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 5 | 2 | 4 | 0 | 2 | 2 | 0 | 1 | 25
  Male | 4 | 6 | 5 | 2 | 4 | 2 | 0 | 2 | 2 | 3 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 5
  Not Hispanic or Latino | 8 | 9 | 10 | 3 | 7 | 2 | 2 | 4 | 1 | 4 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
  Black or African American | 1 | 3 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 11
  White | 7 | 4 | 7 | 3 | 7 | 1 | 1 | 3 | 1 | 2 | 36
  More than one race | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With P.Falciparum Blood Stage Infection
Description: Participants with P. falciparum blood stage infection defined as detection of P. falciparum parasites by qPCR (real time NIH qPCR and sensitive retrospective Laboratory of Malaria Immunology & Vaccinology (LMIV) qPCR) following Sanaria® PfSPZ Challenge (NF54) via direct venous injection (DVI).
Time Frame: 14 days post PfSPZ Challenge injection
Population: Participants who received investigational product
Measure: Number; unit: Participants
Groups:
- Pilot (1b): 1 Dose of 1x10^5 PfSPZ Challenge + Pyrimethamine: Pilot Phase - 1 injection of 1x10^5 sporozoites of PfSPZ Challenge (NF54) with 50mg of pyrimethamine dosed on days 2 and 3 after injection.
- Pilot (1d): 1 Dose of 2x10^5 PfSPZ Challenge + Pyrimethamine: Pilot Phase - 1 injection of 2x10^5 sporozoites of PfSPZ Challenge (NF54) with 50mg of pyrimethamine dosed on days 2 and 3 after injection.
- Main (2a): 3 Doses of 2x10^5 PfSPZ + Pyrimethamine + NF54 CHMI: Main Phase - 3 monthly doses of 2x10^5 sporozoites of PfSPZ Challenge + pyrimethamine on days 2 and 3 post injection + homologous controlled human malaria infection (CHMI) with 3.2x10^3 PfSPZ Challenge (NF54) at 12 weeks after third injection.
- Main (2b): 3 Doses of 2x10^5 PfSPZ + Pyrimethamine + 7G8 CHMI: Main Phase - 3 monthly doses of 2x10^5 sporozoites of PfSPZ Challenge + pyrimethamine on days 2 and 3 post injection + heterologous CHMI with 3.2x10^3 PfSPZ Challenge (7G8) at 12 weeks after third injection.
Arm/Group | Pilot (1a):1 Injection of 5x10^4 PfSPZ Challenge+Pyrimethamine | Pilot (1b): 1 Dose of 1x10^5 PfSPZ Challenge + Pyrimethamine | Pilot (1d): 1 Dose of 2x10^5 PfSPZ Challenge + Pyrimethamine | Main (2a): 3 Doses of 2x10^5 PfSPZ + Pyrimethamine + NF54 CHMI | Main (2b): 3 Doses of 2x10^5 PfSPZ + Pyrimethamine + 7G8 CHMI
Number analyzed (Participants) | 2 | 2 | 4 | 9 | 10
Participants | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Requiring Treatment With Additional Anti-malarial Medication
Description: Incidence of a clinical malaria diagnosis occurring after PfSPZ-Cvac challenge requiring treatment with atovaquone/proguanil (Malarone).
Time Frame: 12 days post PfSPZ Challenge injection
Measure: Number; unit: participants
Groups:
- Main (3): 3 Doses of 2x10^5 PfSPZ + Chloroquine + 7G8 CHMI: Main Phase - 3 monthly doses of 2x10^5 sporozoites of PfSPZ Challenge + weekly chloroquine (1000mg given 2 days prior to injections and 500mg given 5 days post injection and weekly thereafter until 5 days post third injection) + heterologous controlled human malaria infection (CHMI) with 3.2x10^3 PfSPZ Challenge (7G8) at 12 weeks after third injection.
- Pilot (5b): 1 Dose of 2x10^5 PfSPZ Challenge + Chloroquine: Pilot Phase - 1 injection of 2x10^5 sporozoites of PfSPZ Challenge (NF54) with 1000mg of chloroquine (loading dose) 2 days prior to injections and 500mg (maintenance dose) 5 days post injection.
Arm/Group | Main (3): 3 Doses of 2x10^5 PfSPZ + Chloroquine + 7G8 CHMI | Pilot (5a): 1 Injection of 1x10^5 PfSPZ Challenge+Chloroquine | Pilot (5b): 1 Dose of 2x10^5 PfSPZ Challenge + Chloroquine
Number analyzed (Participants) | 10 | 2 | 4
participants | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Local and Systemic Adverse Events (AEs)
Description: Participants who had one or more episodes of related or/and unrelated adverse events (AEs). An AE is defined as any untoward medical occurrence temporarily associated with the subject's participation in research, whether or not considered related or not. Refer to adverse event table for specific AE.
Time Frame: 7 months
Measure: Number; unit: participants
Arm/Group | Pilot (1a):1 Injection of 5x10^4 PfSPZ Challenge+Pyrimethamine | Pilot (1b):1 Injection of 1x10^5 PfSPZ Challenge+Pyrimethamine | Pilot (1d):1 Injection of 2x10^5 PfSPZ Challenge+Pyrimethamine | Main (2a):3 Doses of 2x10^5 PfSPZ Challenge+Pyrimethamine+NF54 | Main (2b):3 Doses of 2x10^5 PfSPZ Challenge+Pyrimethamine+7G8 | Main (3):3 Doses of 2x10^5 PfSPZ Challenge+Chloroquine+7G8 | Pilot (5a): 1 Injection of 1x10^5 PfSPZ Challenge+Chloroquine | Pilot (5b): 1 Injection of 2x10^5 PfSPZ Challenge+Chloroquine
Number analyzed (Participants) | 2 | 2 | 4 | 9 | 10 | 10 | 2 | 4
participants | 2 | 2 | 3 | 8 | 9 | 10 | 2 | 4

4. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Participants who had one or more episodes of serious adverse events (SAEs). SAE is defined as a life-threatening reaction or event that results in death.
Time Frame: 7 months
Measure: Number; unit: participants
Arm/Group | Pilot (1a):1 Injection of 5x10^4 PfSPZ Challenge+Pyrimethamine | Pilot (1b):1 Injection of 1x10^5 PfSPZ Challenge+Pyrimethamine | Pilot (1d):1 Injection of 2x10^5 PfSPZ Challenge+Pyrimethamine | Main (2a):3 Doses of 2x10^5 PfSPZ Challenge+Pyrimethamine+NF54 | Main (2b):3 Doses of 2x10^5 PfSPZ Challenge+Pyrimethamine+7G8 | Main (3):3 Doses of 2x10^5 PfSPZ Challenge+Chloroquine+7G8 | Pilot (5a): 1 Injection of 1x10^5 PfSPZ Challenge+Chloroquine | Pilot (5b): 1 Injection of 2x10^5 PfSPZ Challenge+Chloroquine
Number analyzed (Participants) | 2 | 2 | 4 | 9 | 10 | 10 | 2 | 4
participants | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: Two weeks for pilot phase; four weeks for infectivity controls; seven months for main phase
Arm/Group | Pilot (1a):1 Injection of 5x10^4 PfSPZ Challenge+Pyrimethamine | Pilot (1b):1 Injection of 1x10^5 PfSPZ Challenge+Pyrimethamine | Pilot (1d):1 Injection of 2x10^5 PfSPZ Challenge+Pyrimethamine | Pilot (5a): 1 Injection of 1x10^5 PfSPZ Challenge+Chloroquine | Pilot (5b): 1 Injection of 2x10^5 PfSPZ Challenge+Chloroquine | Main (2a):3 Doses of 2x10^5 PfSPZ Challenge+Pyrimethamine+NF54 | Main (2b):3 Doses of 2x10^5 PfSPZ Challenge+Pyrimethamine+7G8 | Main (3):3 Doses of 2x10^5 PfSPZ Challenge+Chloroquine+7G8 | Main Phase (4a) - Infectivity Control: NF54 (Homologous) CHMI | Main Phase (4b) - Infectivity Control: 7G8 (Heterologous) CHMI
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/4 | 0/2 | 0/4 | 0/9 | 0/10 | 0/10 | 0/4 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/4 | 0/2 | 0/4 | 0/9 | 0/10 | 2/10 | 0/4 | 0/8
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 3/4 | 2/2 | 4/4 | 8/9 | 9/10 | 10/10 | 4/4 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pilot (1a):1 Injection of 5x10^4 PfSPZ Challenge+Pyrimethamine (N=2) | Pilot (1b):1 Injection of 1x10^5 PfSPZ Challenge+Pyrimethamine (N=2) | Pilot (1d):1 Injection of 2x10^5 PfSPZ Challenge+Pyrimethamine (N=4) | Pilot (5a): 1 Injection of 1x10^5 PfSPZ Challenge+Chloroquine (N=2) | Pilot (5b): 1 Injection of 2x10^5 PfSPZ Challenge+Chloroquine (N=4) | Main (2a):3 Doses of 2x10^5 PfSPZ Challenge+Pyrimethamine+NF54 (N=9) | Main (2b):3 Doses of 2x10^5 PfSPZ Challenge+Pyrimethamine+7G8 (N=10) | Main (3):3 Doses of 2x10^5 PfSPZ Challenge+Chloroquine+7G8 (N=10) | Main Phase (4a) - Infectivity Control: NF54 (Homologous) CHMI (N=4) | Main Phase (4b) - Infectivity Control: 7G8 (Heterologous) CHMI (N=8)
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pilot (1a):1 Injection of 5x10^4 PfSPZ Challenge+Pyrimethamine (N=2) | Pilot (1b):1 Injection of 1x10^5 PfSPZ Challenge+Pyrimethamine (N=2) | Pilot (1d):1 Injection of 2x10^5 PfSPZ Challenge+Pyrimethamine (N=4) | Pilot (5a): 1 Injection of 1x10^5 PfSPZ Challenge+Chloroquine (N=2) | Pilot (5b): 1 Injection of 2x10^5 PfSPZ Challenge+Chloroquine (N=4) | Main (2a):3 Doses of 2x10^5 PfSPZ Challenge+Pyrimethamine+NF54 (N=9) | Main (2b):3 Doses of 2x10^5 PfSPZ Challenge+Pyrimethamine+7G8 (N=10) | Main (3):3 Doses of 2x10^5 PfSPZ Challenge+Chloroquine+7G8 (N=10) | Main Phase (4a) - Infectivity Control: NF54 (Homologous) CHMI (N=4) | Main Phase (4b) - Infectivity Control: 7G8 (Heterologous) CHMI (N=8)
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 2 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 4 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 6 | 4 | 4 | 1 | 2
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 2 | 4 | 1 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 1 | 4 | 7 | 6 | 3 | 5
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site induration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 3 | 1 | 3 | 4 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 1 | 1 | 1 | 0 | 3 | 1 | 1 | 1 | 1
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 4 | 8
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 3 | 6 | 4 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Animal scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Heat exhaustion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 4 | 0 | 3
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 3 | 0 | 2
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Smear cervix abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 3 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 3 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 4 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 3 | 3 | 1 | 1 | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 3 | 5 | 5 | 6 | 1 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 1 | 2 | 3 | 3 | 8 | 7 | 3 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0
Alcohol use (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-12): https://cdn.clinicaltrials.gov/large-docs/47/NCT03083847/Prot_SAP_000.pdf